CLINICAL TRIAL: NCT06751602
Title: A Phase 2, Randomized, Placebo-Controlled Study to Evaluate Belumosudil for the Abrogation of Interstitial Fibrosis and Tubular Atrophy in de Novo Kidney Transplant Recipients
Brief Title: Belumosudil for Abrogation of Interstitial Fibrosis and Tubular Atrophy Following Kidney Transplantation
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Caroline Simon, Department of Surgery, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PRO00037984; U1111-1291-6888 (Registry Identifier: WHO International Clinical Trials Registry)
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Rejection Chronic Renal
Keywords: kidney transplantation; RhoA/Rock pathway; interstitial fibrosis/tubular atrophy
MeSH Terms: conditions — Pulmonary Fibrosis | interventions — belumosudil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Belumosudil (Experimental): 200mg/day belumosudil for 12 months
  Interventions: Drug: Belumosudil 200 mg QD
- Placebo (Placebo Comparator): Daily placebo for 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Belumosudil 200 mg QD — Belumosudil 200 mcg oral daily
  Other Names: Rezurock; Belumosudil
  Arms: Belumosudil
Drug: Placebo — Placebo (once daily)
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled trial in de novo kidney transplant patients to determine if the addition of belumosudil (brand name- REZUROCK®) on the background of standard immunosuppression will prevent fibrosis in the kidney transplant. Interstitial expansion is the precursor of interstitial fibrosis and graft loss. The hypothesis underlying the study is that abgrogating the fibrogenic effects of the RhoA pathway with belumosudil will reduce structural damage in transplanted kidneys and possible subsequent transplant failure.

DETAILED DESCRIPTION:
Of the 16,521 adult kidney transplants in 2008, death-censored graft loss occurred in 16% of deceased donor kidneys and 7% of living donor kidneys in the ensuing 5 years and has not largely changed in a decade. A majority of this graft loss is presumed to be from IF/TA, previously termed chronic allograft nephropathy. Various causes of injury to the kidney stimulate inflammatory processes. When the inflammation continues (ie, becomes chronic), changes occur in the kidney structure, specifically in the glomerulus and tubular interstitium which leads to fibrosis and a progressive decline in kidney function.

Interstitial fibrosis and tubular atrophy almost invariably occur together and are present in approximately 45% of early indication kidney biopsies by the first year posttransplant. No risk factors have been identified to predict who will experience IF/TA. Combined, IF/TA contributes to renal graft dysfunction or the decline in kidney function after transplantation and may be a factor in the 20.6% of total grafts lost (including death) by 5 years post-transplant.

Expansion of the interstitial compartment is a major component of IF/TA. Protocol and for-cause biopsies have provided evidence of the worsening of IF/TA with time in kidney transplant recipients and demonstrated a direct relationship between interstitial expansion and renal allograft functional decline and graft failure. Interstitial expansion will be assessed as the overall proportion of cortical tissue area associated with IF/TA.

Previous work has shown that chronic rejection depends on macrophage movement to the graft, which is regulated by actin cytoskeleton controlled by the small GTPase RhoA/Rock pathway. Pharmacologic inhibition or macrophage-specific deletion of RhoA prevents chronic rejection in the rodent cardiac transplantation model, and belumosudil was superior in preventing fibrosis.

Controlling hypertension and prevention and treatment of acute rejection are standard approaches to kidney function preservation in kidney transplant recipients. Additionally, the use of CNI-sparing protocols has been reported with various approaches but data are insufficient to equivocally demonstrate consistently lower IF/TA in the approaches reported to date. Thus, it is important to examine additional approaches for prevention of IF/TA in this population.

This study will test the hypothesis that abrogating the fibrogenic effects of the RhoA pathway with belumosudil would abbrograte IF/TA and that reducing this structural damage in transplanted kidneys would result in improved or preserved kidney function and reduced graft loss.

The purpose of this study is to demonstrate that 200mg/day of belumosudil for 12 months administered to de novo kidney transplant recipients will be safe and to examine the course of IF/TA over a 1-year period by testing the ability of 200mg/day belumosudil for 12 months to abrograte the development of IF/TA in de novo kidney transplant recipients compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Receiving a first or second kidney, except those whose first kidney transplant was lost during year 1 due to rejection or recurrent disease
* Male or female, aged ≥18 to ≤75
* Women of child bearing potential who have a negative serum pregnancy test prior to treatment
* Women of child bearing potential (including perimenopausal women who have had a menstrual period within the previous 1 year) who agree to use 2 forms of effective birth control regimen (at least one of which is a barrier method) throughout the study period and for 6 weeks following the end of the study or the last dose of mycophenolic acid, whichever comes first.
* Sexually active male patients who agree to use effective contraception during treatment of the male patient and for at least 90 days after cessation of treatment with mycophenolic acid.
* Panel of reactive antibodies (PRA) <80% based on the most recent PRA results that are closest to the date of transplant
* Able to take oral medication
* Agreement to adhere to Lifestyle Considerations throughout study duration (refraining from consumption of grapefruit or grapefruit juice; stopping anticoagulation therapy one week prior through one week post-kidney biopsy procedure; agree to follow FDA guidelines regarding contraception while using mycophenolic acid)

Exclusion Criteria:

* Transplantation of any organ other than kidney
* Living donor kidney recipients having a 6-antigen match with their donor or a 0-antigen mismatch
* Planned use of non-calcineurin inhibitor immunosuppression maintenance therapy (eg, belatacept)
* Patients with primary focal segmental glomerulosclerosis
* Recipients of en-bloc kidneys
* Patients who have received or are expected to receive alemtuzumab
* Presence of any donor-specific antibody observed during the current or historical crossmatch assessment
* Presence of primary (or familial) dyslipidemia
* Presence of an increased QTc interval > 480 ms on screening ECG, a history of torsades de pointes, congenital long QT syndrome, bradyarrhythmias, or uncompensated heart failure.
* Patients with a history of CABG, cardiac stent placement, or MI within 1 year prior to enrollment
* Patients taking high intensity statin therapy (ie, atorvastatin 40 or 80mg, rosuvastatin 20-40mg)
* Diagnosed with severe liver disease, including abnormal liver enzymes greater than 3 times the upper limit of normal or total bilirubin greater than 1.5 times the upper limit of normal.
* Diagnosed with any past or present malignancies except squamous or basal cell carcinoma of the skin excised prior to randomization.
* Diagnosed with active acute or chronic infection, or febrile illness, including absolute neutrophil count less than 1.5 K/µL that, in the Principal Investigator's opinion, would impact the patient's safety or any assessments of this study
* Diagnosed with a genetic disease that leads to excessive bleeding (eg, hemophilia A or factor VIII deficiency, hemophilia B or factor IX deficiency, and von Willebrand disease), genetic or acquired disease that leads to excessive clotting (eg, anti-phospholipid syndrome, factor V Leiden thrombophilia, factor II mutation), or a medical condition requiring uninterrupted long-term systemic anticoagulation after transplantation, which would interfere with obtaining biopsies.
* Patient with platelet count less than 50 K/µL.
* Ever diagnosed with Post-Transplant Lymphoproliferative Disorder (PTLD) if a previous kidney transplant was received
* Use of any investigational drug during the 4 weeks prior to enrolling in this study
* Women of child bearing potential who are breastfeeding
* Women of childbearing potential not practicing reliable methods of contraception. Reliable methods for contraception include surgical sterilization (hysterectomy, bilateral tubal ligation), double-barrier method (such as condom and diaphragm). To be considered as post-menopausal and not of childbearing potential, female participants must have experienced 12 consecutive months of amenorrhea.
* Men who are sexually active but do not practice reliable birth control.
* Known allergic reactions to components of REZUROCK®, specifically belumosudil mesylate, microcrystalline cellulose, hypromellose, croscarmellose sodium, colloidal silicon dioxide, magnesium stearate, polyvinyl alcohol, polyethylene glycol, talc, titanium dioxide or yellow iron oxide.
* Any participant whose surgeon expects they will not perform a baseline biopsy pre- or post-reperfusion of the transplanted organ
* Presence of any medical or psychosocial condition, which the investigator believes, would hinder adherence to the study requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Difference in Severe Treatment-Emergent Adverse Events within 12 Months | Time of first dose to 12 months after first dose (study drug/placebo)
  The difference in the proportion of cumulative treatment-emergent adverse events determined to be ≥ grade 3 severity that occur during 12 months from the first dose of belumosudil compared to the placebo group

SECONDARY OUTCOMES:
Proportion of Participants Developing IFTA Progression from Baseline | 12 months after first dose (study drug/placebo)
  The proportion of participants developing progression of interstitial fibrosis/tubular atrophy (IFTA) from baseline assessed on pathology using Banff criteria at 1-year following the first dose of belumosudil or placebo

OTHER OUTCOMES:
Change in Urinary Albumin-to-Creatinine Ratio | 12 months after first dose of study drug or placebo
  Change in participant urinary albumin:creatinine ratio from baseline to 12 months after first dose of study drug or placebo
Urinary Albumin-to-Creatinine Ratio | 12 months after first dose of study drug or placebo
  Participant urinary albumin:creatinine ratio
Change in estimated glomerular filtration rate | 12 months after first dose of study drug or placebo
  Change in estimated glomerular filtration rate (eGFR) from baseline to 12 months after first dose of study drug or placebo
Measured Glomerular Filtration Rate | 12 months after first dose of study drug or placebo
  Measured glomerular filtration rate (mGFR) at 12 months after first dose of study drug or placebo
Graft Loss | 12 months after first dose of study drug or placebo
  Graft loss from causes other than IF/TA or death
Changes in Biomarkers of Fibrosis | 12 months after first dose of study drug or placebo
  Changes in biomarkers of fibrosis (eg, MCP1, Procollagen 3 peptide, BMP-7, TGF-Beta, Wnt4, Cxcl10, Ptx3, MMP-2, CCR2, Notch1) from baseline to 12 months after first dose of belumosudil or placebo
Change in Blood Monocyte Biomarkers | 12 months after first dose of study drug or placebo
  Changes in expression of RhoA, ROCK1, and ADAMTS2 in blood monocytes from baseline to 12 months after first dose of belumosudil or placebo
Biopsy-Proven Acute Rejection | 12 months after first dose of study drug or placebo
  Prevalence of biopsy-proven acute kidney graft rejection within 12 months after first dose of belumosudil or placebo
Banff Score for Interstitial Fibrosis and Tubular Atrophy | 12 months after first dose of study drug or placebo
  Banff score for interstitial fibrosis and tubular atrophy (IFTA) of kidney biopsies at 12 months after first dose of belumosudil or placebo, with the score ranging from i-IFTA0 (no inflammation or less than 10% of cortical parenchyma with IFTA) to i-IFTA3 (inflammation in >50% of cortical parenchyma with IFTA), where i-IFTA3 represents the highest levels for inflammation and IFTA.
iBOX Score | 6 and 12 months after kidney transplantation
  Difference between belumosudil and placebo in mean iBOX score (iBOX kidney transplant risk prediction tool, -7 to +1; negative values indicate better score) at 6 months and 1 year post-transplant

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist Research Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen W, Chen W, Chen S, Uosef A, Ghobrial RM, Kloc M. Fingolimod (FTY720) prevents chronic rejection of rodent cardiac allografts through inhibition of the RhoA pathway. Transpl Immunol. 2021 Apr;65:101347. doi: 10.1016/j.trim.2020.101347. Epub 2020 Oct 24. PMID 33131698
- [Background] Chen W, Chen S, Chen W, Li XC, Ghobrial RM, Kloc M. Screening RhoA/ROCK inhibitors for the ability to prevent chronic rejection of mouse cardiac allografts. Transpl Immunol. 2018 Oct;50:15-25. doi: 10.1016/j.trim.2018.06.002. Epub 2018 Jun 6. PMID 29885441
- [Background] Subuddhi A, Uosef A, Zou D, Ubelaker HV, Ghobrial RM, Kloc M. Comparative transcriptome profile of mouse macrophages treated with the RhoA/Rock pathway inhibitors Y27632, Fingolimod (Gilenya), and Rezurock (Belumosudil, SLx-2119). Int Immunopharmacol. 2023 May;118:110017. doi: 10.1016/j.intimp.2023.110017. Epub 2023 Mar 15. PMID 36931169